CLINICAL TRIAL: NCT01050192
Title: The Nutritional Content of Breast Milk From Mothers of Premature Neonates During the First 28 Days of Life
Brief Title: Nutritional Content of Breast Milk From Mothers of Premies
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Pediatrix (Other)
Collaborators: Prolacta Bioscience (Industry)
Responsible Party: Principal Investigator, Amy Kelleher, Director Clinical Trial Operations, Pediatrix
Other Study IDs: Pro0001271
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Prematurity; Nutrition
Keywords: Prematurity; Nutrition; Breast Feeding
MeSH Terms: conditions — Premature Birth; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the correlation, if any, between the nutritional content of breast milk pumped by the mothers of very low birth weight (VLBW) infants in the neonatal intensive care unit (NICU) and the nutritional value they are actually receiving in a 24 hour period, since as a practical matter, these may not be the same.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of infants with a gestational age <=30 weeks in the NICU who are supplying their own breast milk for use by their baby
* Reasonable likelihood of survival of infant to 28 days
* Infant on/ready for oral feeding by DOL 7 days
* Willing to provide breast milk for their baby
* Able to produce at least 7mL breast milk per feeding
* Willing to abide by requirements of the study protocol
* Documentation of informed consent

Exclusion Criteria:

* Unable to provide at least 7mL breast milk per feeding
* Medically unsuitable to provide breast milk to her baby
* Maternal age <18 years of age

Ages: 23 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Neonatal Intensive Care Unit
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To determine the correlation, if any, between the nutritional content of breast milk pumped by the mothers of VLBW infants in the NICU and the nutritional value they are actually receiving in a 24 hour period. | 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Reese Clark, MD, Principal Investigator — Greenville Memorial Hospital
Locations (1):
- Greenville Memorial Hospital, Greenville, South Carolina, United States